CLINICAL TRIAL: NCT06971510
Title: The Effectiveness of Robotic Exoskeleton on Sensori-motor Performance in Subjects With Incomplete Spinal Cord Injury: A Functional Near-Infrared Spectroscopy Study
Brief Title: Exoskeleton Training on Balance Control and Turning in Ambulation in Individuals With Incomplete Spinal Cord Injury
Acronym: iSCI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Collaborators: The Affiliated BenQ Hospital of Nanjing Medical University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HE-OT2021/16
Record Dates: First submitted 2024-05-28; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2024-12

CONDITIONS: Spinal Cord Injuries
Keywords: Exoskeleton training; Balance; Turning; Gait; Neuroplasticity; Quality of life
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: 1) Exoskeleton training group, 2) conventional training group; 3) usual care group
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Exoskeleton Training Group (Experimental): EksoNR robotic training includes 10 min warm-up, and 5 min cool down (2x/wk, 12 weeks, 24 sessions), minimum 300 steps per session after the third session. The 45 min training excludes set-up/donning/doffing time and includes standing/up time, walking time, and seated rest breaks. The EksoNR training includes weight shift, stepping, straight walking with symmetry gait pattern, and turning with asymmetry gait pattern.
  Interventions: Device: Exoskeleton Training
- Conventional Training Group (Active Comparator): Participants in this group will receive 24-session conventional physical therapy (2x/wk, 12 weeks). Each session lasts 60 minutes, including 10 min warm-up, and 5 min cool-down. Conventional training includes mobilization exercises, strengthening exercises, and balance and gait training. The sessions will be supervised by a trained physiotherapist who will provide guidance and cues to the participants throughout. EksoNR training sessions will be provided after the completion of all the assessments.
  Interventions: Other: Conventional Physical Therapy
- Usual Care Group (No Intervention): Participants in this group continue with daily activities as normal over 12 weeks. No new gait training, mobility therapy, or new medications related to the condition under study, will be commenced during the study period. Participants in this group come to the study sites for evaluations at baseline, 6 weeks, 12 weeks, and one-month follow-up. EksoNR training sessions will be provided after the completion of all the assessments.

INTERVENTIONS:
Device: Exoskeleton Training — Using EksoNR to train balance control and walking and turning abilities in patients with incomplete spinal cord injury.
  Arms: Exoskeleton Training Group
Other: Conventional Physical Therapy — Using conventional physical therapy methods to train the balance control and walking and turning abilities in patients with incomplete spinal cord injury.
  Arms: Conventional Training Group

SUMMARY:
This study investigates the impact of exoskeleton training on individuals with incomplete spinal cord injury (iSCI). Investigators focus on assessing how the use of the exoskeleton influences balance control and turning during ambulation and quality of life in this population. The study mainly involves interventions with participants utilizing exoskeleton devices to explore the influence on mobility, stability, and neuroplasticity, providing new insights into the potential benefits of exoskeleton training for individuals with incomplete spinal cord injuries.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) poses profound challenges to individuals, disrupting complex neural pathways responsible for motor and sensory functions. Across a spectrum of impairments, the ability to navigate and maneuver during walking, particularly turning, is a significant obstacle for patients with incomplete SCI (iSCI). Despite advances in rehabilitation strategies, turning-while-walking remains a biomechanically demanding task that is often overlooked in traditional interventions that focus primarily on linear gait training.

Turning-while-walking requires coordinated movements of the head, trunk, pelvis, and limbs. Disruption of sensory pathways and impairment of motor control after iSCI complicates this complex process, resulting in impaired balance, increased risk of falls, and decreased quality of life. While traditional rehabilitation methods strive to address these challenges, they often fail to target the specific complexities of turning dynamics.

Robotic exoskeletons are wearable devices designed to enhance mobility for iSCI patients. These innovative technologies are expected to enhance sensorimotor performance by providing external support, promoting gait symmetry, and promoting neuroplasticity through intensive training. Exoskeleton-assisted therapy has the potential not only to restore physical function, but also to promote psychosocial well-being, allowing individuals to participate more fully in daily activities and social interactions.

However, despite the growing body of research demonstrating the benefits of exoskeleton training, its efficacy in improving turning-while-walking performance among individuals with iSCI remains uncertain. Furthermore, the neurological mechanisms underlying the response to exoskeleton training in this population warrant deeper investigation.

This study aims to elucidate the effectiveness of a robotic exoskeleton on sensorimotor performance in subjects with iSCI. By filling gaps in the existing literature through rigorous methodology and comprehensive evaluation, investigators strive to provide valuable insights into the potential of exoskeleton-assisted therapy to optimize rehabilitation outcomes and improve the lives of iSCI survivors. Through a multidimensional approach encompassing both physical and psychosocial domains, this research seeks to pave the way for more tailored and effective interventions in SCI rehabilitation, ultimately fostering greater independence and well-being for those affected by this debilitating condition.

The objective of the cluster randomized controlled trial is to investigate the effectiveness of exoskeleton training specifically on turning-while-walking performance, balance control, gait function, muscle strength, spasticity, quality of life, self-efficacy, and fall incidence in people with iSCI. Moreover, the study will also explore how exoskeleton training may promote neuroplasticity and its relationship with ambulatory function and balance control changes in people with iSCI. The three centers will serve as distinct clusters and will be randomized into three groups: 1) Exoskeleton Training Group (ETG), 2) Conventional Exercise Group (CEG), and 3) Usual Care Control Group (UCG). The ETG and CTG will undergo 24 training sessions over 12 weeks respectively, and the UCG will receive standard care.

Assessments will be conducted at baseline, midpoint (Week 6), post-intervention (Week 12), and one-month post-intervention to evaluate outcomes such as turning-while-walking performance, balance control, gait performance, muscle strength, spasticity, self-efficacy, fall incidence, and quality of life. Additionally, cortical activity will be measured to explore changes in neural pathways and their correlation with turning performance and balance control during ambulation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years
2. Traumatic or non-traumatic SCI, > 6 months since SCI onset Motor incomplete SCI (American Spinal Injury Association Impairment Scale, AIS C and D), neurologic level of injury (NLI) between C1-L2 (inclusive), as determined by the International Standards for Neurological Classification of SCI (ISNCSCI)
3. Able to walk with or without walking aid independently for at least 2 meters
4. No current or history of other neurological conditions
5. Community-dwelling or living in a rehabilitation facility
6. Medically stable for full weight-bearing locomotor training including 15-minute standing frame trial to assess standing tolerance
7. Weigh 220 pounds (100 kg) or less (exoskeleton equipment requirement)
8. Between approximately 1.5 m and 1.9 m (5'0" and 6'4") tall (exoskeleton equipment requirement)
9. Standing hip width of approximately 45 cm (18") or less (exoskeleton equipment requirement)
10. Sufficient range of motion (ROM) to achieve a normal, reciprocal gait pattern, and normal sit-to-stand transitions.

    Hip extension greater than or equal to 5-degree Knee extension greater than or equal to 5-degree Ankle dorsiflexion greater than or equal to 0-degree
11. Sufficient upper extremity strength to use a front wheeled walker by manual muscle testing (minimum triceps strength bilaterally of 3/5 of Oxford Scale, shoulder abduction and flexion/extension 4/5 of Oxford Scale)

Exclusion Criteria:

1. AIS-A SCI or AIS-B SCI
2. Have been trained in exoskeleton or other robotic device for locomotor training within the past 4 months except for one or two training/demonstration sessions
3. Currently involved in another intervention study
4. Any medical issue that precludes full weight-bearing locomotor training including but not limited to:

   Spinal instability (or spinal orthotic unless cleared by physician) Acute deep vein thrombosis (DVT) with activity restrictions Severe, recurrent autonomic dysreflexia (AD) requiring medical intervention Heterotopic ossification (HO) in the lower extremities resulting in ROM restrictions at the hips or knees Two or more pathological fractures in the last 48 months in a major weight-bearing bone (femur or tibia) in the lower extremity Hip subluxation (x-rays will be obtained for individuals injured prior to 10 years of age)
5. Any medical issue that would affect participant safety either due to cognitive deficits/impulsivity, intolerance to mild exercise, or other factors
6. Any issue that would confound results such as a concurrent neurological injury or disorder (other than SCI) or other factors
7. Skin integrity issues in areas that contact the device (including abdominal ostomies) or that would prohibit sitting
8. Pregnancy
9. Participants who do not meet the exoskeleton equipment requirements
10. Modified Ashworth Scale (MAS) = 4 in the majority of lower extremity joints (e.g. greater than or equal to four joint movements in bilateral lower extremities when testing hip flexion/extension, knee flexion/extension, ankle dorsi/plantar flexion)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Duration of a turn | baseline, session 12 (6 Weeks), session 24 (12 Weeks), 1-month follow-up
  The participants are asked to walk a straight line of 1 meter, execute a 180-degree turn, and return to the starting position as quickly and safely as possible. Participants have the flexibility to use any necessary walking aids and wear their ankle-foot orthotics as needed. A turn is defined as starting and completing a 180-degree change in walking direction at a marked turn spot on the floor. The start of the turn is determined as the last foot contact prior to the inanition of the direction change. The end of the turn is determined as the last foot contact when both feet turn in the backward direction. Two tripod-mounted video cameras are placed in sagittal plane and frontal plane respectively.
  An assessor will view the videotapes of the turn by using a video-cassette player. The duration of a turn will be extracted and computed averages of three trials on each side.
Number of steps to a turn | baseline, session 12 (6 Weeks), session 24 (12 Weeks), 1-month follow-up
  The participants are asked to walk a straight line of 1 meter, execute a 180-degree turn, and return to the starting position as quickly and safely as possible. Participants have the flexibility to use any necessary walking aids and wear their ankle-foot orthotics as needed. A turn is defined as starting and completing a 180-degree change in walking direction at a marked turn spot on the floor. The start of the turn is determined as the last foot contact prior to the inanition of the direction change. The end of the turn is determined as the last foot contact when both feet turn in the backward direction. Two tripod-mounted video cameras are placed in sagittal plane and frontal plane respectively.
  An assessor will view the videotapes of the turn by using a video-cassette player. The number of steps to a turn will be extracted and computed averages of three trials on each side.

SECONDARY OUTCOMES:
Limits of Stability (LOS) | baseline, session 12 (6 Weeks), session 24 (12 Weeks), 1-month follow-up
  The Limits of Stability (LOS) test assesses dynamic balance using the Biodex Medical System. Participants stand on a stable platform (level 12) with feet positioned to maintain balance over the center. The test measures the time and accuracy as participants lean to intercept eight targets displayed at 45° intervals around a central point representing their center of pressure. Each target is randomly highlighted, and participants must reach each target as quickly and accurately as possible, returning to the center between attempts. Targets are set at 50% of the LOS based on participant height, and practice trials precede the main test. Participants can use handles briefly for balance recovery, but excessive reliance on them will terminate the test. Key outcomes include the time taken to reach targets and directional control, calculated as a percentage of accuracy. Three trials are recorded, and averaged values are used for statistical analysis.
Modified Clinical Test of Sensory Integration and Balance (m-CTSIB) | baseline, session 12 (6 Weeks), session 24 (12 Weeks), 1-month follow-up
  The Modified Clinical Test of Sensory Integration and Balance (m-CTSIB) is assessed using the Biodex Balance SD (Biodex Medical System, Inc., New York, USA). This test evaluates the effects of sensory integration on standing balance across four conditions: eyes open on a firm surface, eyes closed on a firm surface, eyes open on a foam surface, and eyes closed on a foam surface. Each condition lasts 30 seconds, with a minimum 10-second rest period between trials as needed. Participants complete practice trials prior to the test trials, and the order of testing is randomized to minimize learning effects. Balance performance is quantified using the Sway Index (SI), where a higher SI indicates greater instability. The SI is recorded for each condition, along with a final overall SI. Three trials are conducted for each condition, and averages of the individual conditions and overall SI are calculated for data analysis.
Muscle strength | baseline, session 12 (6 Weeks), session 24 (12 Weeks), 1-month follow-up
  A hand-held dynamometer will assess the strength of bilateral lower limbs (hip flexors, extensors, abductors, adductors, knee flexors, extensors, ankle dorsiflexors, and plantarflexors) in a lying position, as well as trunk muscles (flexors, extensors, and rotators) in a sitting position. Each muscle strength test will be performed three times, and the averaged values will be used for data analysis.
Modified Ashworth Scale (MAS) | baseline, session 12 (6 Weeks), session 24 (12 Weeks), 1-month follow-up
  The Modified Ashworth Scale (MAS) assesses spasticity in various muscles bilaterally, including hip flexors, extensors, adductors, knee flexors, extensors, and ankle dorsiflexors and plantarflexors. Scores range from 0 to 5, where 0 indicates no spasticity and 5 indicates severe spasticity. Higher scores reflect worse outcomes in terms of spasticity levels.
Modified Functional Reaching Test (MFRT) | baseline, session 12 (6 Weeks), session 24 (12 Weeks), 1-month follow-up
  The Modified Functional Reaching Test (MFRT) will assess participants' balance while seated on a chair without back or arm support. A yardstick will be positioned at the level of the acromion, with participants' feet flat on the ground. Starting with one shoulder flexed to 90 degrees, the ulnar styloid process will be the anatomical landmark for measuring reach. Participants will reach forward, backward, and laterally as far as possible without trunk rotation, with a research team member providing safety support. The maximum distance reached in centimeters for each direction will be recorded. Each direction will be tested three times, and the average value for each direction will be used for data analysis.
Berg Balance Scale (BBS) | baseline, session 12 (6 Weeks), session 24 (12 Weeks), 1-month follow-up
  The Berg Balance Scale (BBS) assesses functional mobility and balance through 14 tasks evaluating both static and dynamic balance. Each task is scored on a 5-point ordinal scale from 0 to 4, with 0 indicating the lowest level of function and 4 the highest. The total score ranges from 0 to 56, with higher scores indicating better balance and functional mobility. Scoring is based on the participant's ability to meet specific time or distance requirements and to perform tasks independently. Participants wear their usual shoes and any necessary orthotics during testing, but they are not allowed to use walking assistive devices.
The Timed Up and Go Test (TUGT) | baseline, session 12 (6 Weeks), session 24 (12 Weeks), 1-month follow-up
  The Timed Up and Go Test (TUGT) is a test that involves various mobility activities that are common in daily life. When the test started, the subject should stand up from a seated position, walk straight forward for three meters, turn around, walk back to the starting position, and then sit down. The test will be repeated three times. The average time taken to complete the whole process will be used for data analysis.
10 Meter Walk Test (10MWT) | baseline, session 12 (6 Weeks), session 24 (12 Weeks), 1-month follow-up
  10 Meter Walk Test (10MWT) is used to assess the walking speed of participants. Participants will be asked to walk at their maximum walking speed, with their usual walking aid if needed, for 10 meters. The initial and last two meters of the test will be allowed for acceleration and deceleration. The time required to walk for the intermediate six meters will be recorded. The average of three trials will be used for data analysis.
Walking index for spinal cord injury (WISCI II) | baseline, session 12 (6 Weeks), session 24 (12 Weeks), 1-month follow-up
  The Walking Index for Spinal Cord Injury II (WISCI II) is used to classify participants' level of walking independence and the use of assistive devices or braces. This 20-item scale ranges from 0, indicating that the participant is unable to walk, to 20, which signifies that the participant can ambulate 10 meters without assistance, devices, or braces. Higher scores reflect greater walking independence.
Fall incidence | baseline, session 12 (6 Weeks), session 24 (12 Weeks), 1-month follow-up
  Fall history will be assessed with a semi-structured interview by asking the participants about occurrence and frequency of falls during the last 12 month. A fall is defined as any fall, including a slip or a trip, in which the participant came to rest on the floor, ground, or on a lower level. All falls are recorded through weekly self-reports by participants, during the intervention and follow-up.
The 36-Item Short Form Health Survey (SF-36) | baseline, session 12 (6 Weeks), session 24 (12 Weeks), 1-month follow-up
  The 36-Item Short Form Health Survey (SF-36) will be administered to participants to assess their quality of life. Participants will complete the survey, which consists of 36 questions covering eight health dimensions: physical functioning (PF), social functioning (SF), role physical (RP), role emotional (RE), mental health (MH), vitality (VT), bodily pain (BP), and general health (GH) perceptions. Responses will be scored on a standard 0 to 100 scale, where higher scores indicate better health-related quality of life (Forchheim et al., 2004). Data analysis will involve calculating overall total scores as well as individual scores for each dimension.
Falls Efficacy Scale International (FES-I) | baseline, session 12 (6 Weeks), session 24 (12 Weeks), 1-month follow-up
  The Falls Efficacy Scale International (FES-I) is utilized to assess participants' concerns about falling during various daily activities. This scale comprises 16 items, each rated on a 4-point Likert scale from 1 (not at all concerned) to 4 (very concerned), resulting in a total score ranging from 16 (lowest concern) to 64 (highest concern), with higher scores indicating greater concern about falling. Thus, higher scores represent a worse outcome in terms of fall-related anxiety.
Physical Activity Scale for Persons with Physical Disabilities (PASIPD) | baseline, session 12 (6 Weeks), session 24 (12 Weeks), 1-month follow-up
  The Physical Activity Scale for Persons with Physical Disabilities (PASIPD) is used to assess physical activity participation. his 13-item questionnaire quantifies the level of physical activity across leisure, household, and occupational activities over the past seven days. A total score is calculated for data analysis, with potential scores ranging from 0 (no physical activity) to higher values reflecting greater levels of activity.

OTHER OUTCOMES:
Brain hemoglobin concentration | baseline and session 24 (12 Weeks)
  Four participants in the exoskeleton training group will undergo additional measurements of brain hemoglobin concentration using functional near-infrared spectroscopy (fNIRS). The changes in concentration of oxyhemoglobin (HbO2) and deoxyhemoglobin (HbR) will be measured under 3 conditions: 1-minute static standing; 5-meter walking-while-turning overground without exoskeleton; 5-meter walking-while-turning overground within exoskeleton. Five trials will be recorded for each condition. Data will be processed and analyzed in MATLAB using the SPM toolbox.

CONTACTS AND LOCATIONS:
Overall Officials: William WN Tsang, PhD, Study Chair — Department of Physiotherapy, School of Nursing and Health Studies, Hong Kong Metropolitan University
Locations (3):
- China (3):
  - Changzhou Sunshine Rehabilitation hospital, Changzhou, Jiangsu
  - Rehabilitation Medicine Department, The Affiliated BenQ Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Hong Kong Metropolitan University, Hong Kong

IPD SHARING:
Plan to Share IPD: No